CLINICAL TRIAL: NCT04184856
Title: What is Driving the Binge in Binge Eating Disorder? Variability in Brain Response to Reward and the Escalation of Consumption
Brief Title: Binges and Neural Variability
Acronym: BEDVAR
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Else Kröner Fresenius Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: BEDVAR
Record Dates: First submitted 2019-10-29; First posted 2019-12-04 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-04

CONDITIONS: Binge-Eating Disorder
Keywords: reward sensitivity; neuroimaging; variability; ecological momentary assessment (EMA)
MeSH Terms: conditions — Binge-Eating Disorder | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Binge eating disorder (BED) patients: Individuals with BED diagnosis.
  Interventions: Diagnostic Test: fMRI
- non-BED controls: Individuals that do not experience binges
  Interventions: Diagnostic Test: fMRI
- subsyndromal BED controls: individuals that experience binges but do not fulfill the requirements for BED diagnosis.
  Interventions: Diagnostic Test: fMRI

INTERVENTIONS:
Diagnostic Test: fMRI — (Imaging while) performing reward related tasks.

SUMMARY:
People who suffer from binge eating disorder experience recurrent episodes of binge eating.During these episodes, they consume an unusually large amount of food in a short amount of time and experience loss of control over eating. However, why such binge eating episodes occur is still largely unknown. This makes it difficult to develop targeted treatments. In this project, the experimenters are investigating the brain mechanisms that give rise to the disorder. They hypothesize that the binge eating episodes are due to an increased variability in reward processing, which they will assess repeatedly over days. They will test this hypothesis using mathematical models based on behavioural and MRI measurements that are related to the processing of rewards.

ELIGIBILITY:
Inclusion Criteria:

* Binge eating disorder diagnosis
* Subsyndromal binge eating (control)

Exclusion Criteria:

* high risk of suicide
* co-occurring psychotic, bi-polar disorders, alcohol/substance dependence within the past six months
* lack of capacity for consent
* medical disorders that would affect weight and ability to participate
* insufficient German language skills (assessment will be in German)
* taking medication that would affect weight
* MRI exclusion criteria
* irremovable metal attached to the body (e.g. piercings)
* irremovable medical devices (e.g. pacemakers)
* any trauma or surgery which may have left ferromagnetic material in the body
* large tattoos
* pregnancy
* claustrophobia

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The control group will consist of residents of the general area around Tübingen, Germany.
  BED patients will be recruited mainly from the outpatient clinic of the Department of Clinical Psychology of Tübingen, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Variability in blood-oxygen-level dependent (BOLD) signalling in the NAcc during effort allocation task | 100 min
  Variability of BOLD signal in the nucleus accumbens (NAcc) over time and between trials while performing an effort allocation task. The signal is measured through functional magnetic resonance imaging (fMRI) and variability is determined through model residuals.
Trial-to-trial variability in reward seeking in an effort allocation task | 40 min
  Variability of performance is an intra-individual measure, that is defined by the residuals of a linear mixed effects model of trial-to-trial performance on the effort allocation task.
Variability in BOLD signalling in the NAcc for food-cue reactivity | 15
  Variability of BOLD signal in the NAcc between blocks of food pictures. The signal is measured through fMRI and variability is determined through model residuals.

SECONDARY OUTCOMES:
Variability in BOLD signalling in the NAcc during non-food-cue reactivity | 5
  Variability of BOLD signal in the NAcc between blocks of non-food pictures. The signal is measured through fMRI and variability is determined through model residuals.

CONTACTS AND LOCATIONS:
Overall Officials: Nils B Kroemer, Dr, Principal Investigator — University Hospital Tuebingen
Locations (1):
- Psychological Institute, University of Tübingen, Tübingen, Deutschland (deu), Germany